CLINICAL TRIAL: NCT02989272
Title: Effect of Pre-treatment With Magnesium Sulfate on the Duration of Deep Neuromuscular Blockade With Rocuronium: Random and Double-blind Clinical Study
Brief Title: Effect of Pre-treatment With Magnesium Sulfate on the Duration of Deep Neuromuscular Blockade With Rocuronium
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Federal de Bonsucesso (Other)
Responsible Party: Principal Investigator, angelo jorge queiroz rangel micuci, Doctor Anesthesiologist, Hospital Federal de Bonsucesso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HFBonsucesso
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Magnesium Sulfate; Neuromuscular Blockade; Rocuronium; Deep Neuromuscular Blockade
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline group (Placebo Comparator): Control group (30 patients), who will receive Treatment by venous infusion of saline solution
  Interventions: Other: saline group
- Sulfate group (Experimental): magnesium group (30 patients) who will receive pre- Venous infusion of magnesium sulphate 60 mg / kg
  Interventions: Drug: Sulfate, Magnesium

INTERVENTIONS:
Drug: Sulfate, Magnesium — magnesium group (30 patients) who will receive pretreatment by intravenous infusion of magnesium sulfate 60 mg / kg
  Arms: Sulfate group
Other: saline group — saline group (30 patients) who will receive pretreatment by saline solution
  Arms: saline group

SUMMARY:
It is a prospective, comparative, randomized, double-blind clinical trial whose hypothesis is that pre-treatment with magnesium sulfate, due to its action at the neuromuscular junction,potentiate the duration of deep neuromuscular block following rocuronium curarization in patients undergoing general anesthesia. Magnesium sulphate has gained prominence as an adjuvant drug in anesthesia. Its use is associated with potentiation of neuromuscular blockade among other functions.

The deep neuromuscular block is defined as the one obtained by the absence of response to the sequence of four Stimuli and the presence of one or more simple stimuli in post-tetanic counts . There is no literature description of the role of magnesium sulphate in Duration of the deep neuromuscular block obtained after the muscle relaxation of patients with rocuronium This study is justified because extending the clinical duration of neuromuscular blockers may translate into gains for surgeries that require deep and long-lasting muscle relaxation as in laparoscopic and robotic surgeries. This block allows lower inflation pressures of the pneumoperitoneum to be obtained, as a result, there is a lower inflammatory and cardiorespiratory repercussion for the patient

DETAILED DESCRIPTION:
Patients will be selected from those who use the General Surgery Service of the Federal Hospital of Bonsucesso for medical indication or own will, obeying the inclusion and exclusion criteria. After signing the informed consent, they will be evaluated clinically and laboratorially, according to the routine of preoperative exams and pre-anesthetic outpatient evaluation. Patients will be allocated to one of two groups: control group (30 patients), who will receive pretreatment by venous infusion of saline solution; And magnesium group (30 patients) who will receive pretreatment by intravenous infusion of magnesium sulfate 60 mg / kg according to the random number sequence generated electronically through the QuickCalcs program (GraphPad Software, San Diego, CA) Because it is a double-blind study, both the researcher and the patient will not know which of the groups will be studied.

The principal investigator will be responsible for the delivery of sealed envelope containing the sequence of cases allocated in each of the groups to another anesthesiologist who will prepare the solution (saline or magnesium sulphate) and will record in a specific file in which group the volunteer was Allocated. Again the envelope will be sealed for tabulation later, without the knowledge of the researcher. The same principal investigator will be in charge of the measurement and recording of the data collected.

ELIGIBILITY:
Inclusion Criteria:

* Physical State American Society of Anesthesiologists (ASA) I, II and III; Body mass index between 18.5 and 24.9;Otorhinolaryngological surgeries

Exclusion Criteria:

Refusal to participate in the study;

* Pregnancy or suspected pregnancy; Neuromuscular diseases, renal or hepatic impairment;
* Hepatic dysfunction;
* History or predictors of difficult airway; Hypermagnesemia (Mg> 2.5 mEq / L);
* Hypomagnesemia (Mg <1.7 mEq / L);
* Use of furosemide, aminoglycosides, aminophylline, azathioprine; Cyclophosphamide, anti-inflammatories and magnesium;
* Allergy to the drugs used in the study;
* Participants from other clinical studies.
* Emergency surgeries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
duration of deep neuromuscular block | perioperative
  To determine the duration of deep neuromuscular block following a single dose of rocuronium

SECONDARY OUTCOMES:
onset time and recovery time of rocuronium | perioperative- until 48h
  to determine the pharmacodynamic parameters of rocuronium
residual neuromuscular block in PACU | 6h
  Evaluate the eventual occurrence of residual neuromuscular block in PACU
evolution of the height of T1 | perioperative- until 48h
  Record the evolution of the height of T1
postoperative pain | perioperative- until 48h
  Evaluate postoperative pain with questionnaire and visual scale of pain
episodes of nausea and vomiting and treatment of surgery to discharge | perioperative- until 48h
  Assess the frequency of individual episodes of nausea and vomiting and treatment during the period from the end of surgery to discharge
frequency of pain or unpleasant sensation | perioperative- until 48h
  Evaluate frequency of pain or unpleasant sensation during the infusion of the studied solutions

CONTACTS AND LOCATIONS:
Overall Officials: Nubia V Figueiredo, master, Study Director — Universidade Federal do Rio de Janeiro; Ismar L Cavalcanti, master, Study Director — Federal Fluminense University; Angelo Jorge Q R Micuci, doctor anesthesiology, Principal Investigator — Hospital federal of Bonsucesso
Locations (1):
- Bonsucesso Federal Hospital, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Queiroz Rangel Micuci AJ, Vercosa N, Filho PAG, de Boer HD, Barbosa DD, Cavalcanti IL. Effect of pretreatment with magnesium sulphate on the duration of intense and deep neuromuscular blockade with rocuronium: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jul;36(7):502-508. doi: 10.1097/EJA.0000000000001003. PMID 30985540